CLINICAL TRIAL: NCT06515288
Title: The Effect of a School-based Nutrition Intervention to Promote Healthy Eating Behaviour Among Adolescents in Indonesia - a Cluster Randomized Pilot Study
Brief Title: Nutrition Goes to School: a School-based Nutrition Intervention to Promote Healthy Eating Behaviour Among Adolescents
Acronym: ESTEEM-NGTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SEAMEO Regional Centre for Food and Nutrition (Other)
Collaborators: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Indah Widyahening, Professor, SEAMEO Regional Centre for Food and Nutrition
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ESTEEM NGTS
Record Dates: First submitted 2024-07-16; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Obesity, Adolescent
Keywords: School-based intervention; obesity; adolescent; prevention; nutrition
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Five intervention schools and five control schools will be selected from five different municipalities in Jakarta, with each school having a minimum of 100 students (grade 10-11; 15-17 years old). First, recruitment will be based on the discussion with the local education office at the provincial level and ask for a list of schools considering eligibility criteria. Two schools in each municipality with comparable characteristics will be selected, and then each pair will be randomized to become either the intervention or the control group. Second, selected schools will be invited to participate in the study. The intervention group will receive baseline educational intervention (Nutrition Education Capacity Building for Teachers and Management) and all components of the NGTS program. While the control group will receive only the baseline educational intervention. The baseline educational intervention will be conducted in 5 days through face-to-face delivery training mode.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention schools (Experimental): The intervention group will receive baseline educational intervention (Nutrition Education Capacity Building for Teachers and Management) and all components of the Nutrition Goes to School (NGTS) program.
  Interventions: Behavioral: Nutrition Goes To School (NGTS) Program Intervention Package; Behavioral: Nutrition Education Capacity Building for Teachers and Management
- Control schools (No Intervention): The control group receive no specific intervention other than current school health program conducted by the local public health centers (puskesmas).

INTERVENTIONS:
Behavioral: Nutrition Goes To School (NGTS) Program Intervention Package — The NGTS Program intervention package in this project consists of four components:
  1. A comprehensive Nutrition Education to improve healthy eating, physical activity, and hygiene-sanitation practices.
     This is a weekly interactive and fun nutrition and health promotion with different kinds of activities.
  2. Healthy School Canteen to improve the availability of healthy food in school. This is an effort to strengthen the school canteen referring to the 4 Pillars of a Healthy School Canteen, including School Commitment and Management, Human Resources, Facilities and Infrastructure, and Food Quality.
  3. School Garden. This is a gardening activity as a form of school garden as a media for nutrition education, character building, and contribute to supply vegetables during cooking class sessions in school.
  4. Entrepreneurship nutrition. Entrepreneurship nutrition aims to foster entrepreneurial potential and skills among school members in providing healthy food at school.
  Arms: Intervention schools
Behavioral: Nutrition Education Capacity Building for Teachers and Management — The intervention schools will receive Nutrition Education Capacity Building for Teachers and School Management, before the above four NGTS components is implemented in the respective school. Three representatives from each school will be invited to attend a 5-day training that include knowledge on adolescent nutrition and health issues, as well as skills in implementing the NGTS Program.
  Arms: Intervention schools

SUMMARY:
The goal of this cluster randomized controlled pilot trial is to assess the feasibility and effect of a school-based nutrition intervention program called "Nutrition Goes to School" (NGTS) in improving a healthy diet and physical activities as part of the prevention and management of obesity among adolescents in urban Indonesia. The main questions it aims to answer concern the feasibility of the NGTS multi-component school-based nutrition intervention model in selected secondary schools in an urban setting to inform the design of the future effectiveness study. Additionally, it aims to evaluate the effect of the school-based nutrition intervention in the healthy eating knowledge and behavior (fruit and vegetable consumption, energy-dense nutrient poor food, and sugary beverages consumption, as measured by food frequency questionnaire) and physical activities as well as its effect on nutrition status (body mass index, mid-upper arm circumference [MUAC] and waist circumference). The intervention components consist of nutrition education to school communities (teachers, management, students and parents), healthy school canteen, school garden, hygiene and sanitation promotion of the school environment and obesogenic environment control, and promotion of physical activities among students. Five secondary schools in Jakarta will be randomly assigned to receive the intervention for 6 months, and five other schools will serve as the control group.

DETAILED DESCRIPTION:
A program which is called "Nutrition Goes to School" (NGTS) has been initiated by the Southeast Asian Ministers of Education Organization Regional Centre for Food and Nutrition (SEAMEO RECFON) in 2016 to improve the health of the children through implementation of nutrition good practices at schools.The program was started by providing training to school teachers about nutrition and continuously improved until it currently includes multiple components consisting of school readiness survey, healthy school canteen, school garden for nutrition literacy, nutrition education, school hygiene and sanitation promotion and promotion of physical activities at school.

Since its initiation in mid-2016, some schools from primary to secondary level in several provinces in Indonesia have been trained in the implementation of some components of the program. However, since the program was developed gradually and schools' participation is on voluntary basis, no schools participated in the training currently implement the whole components, no standard protocol for the activities was implemented and an impact assessment is yet to been conducted. SEAMEO RECFON is one of the regional organizations under the Ministry of Education in Association of South-east Asian Nations (ASEAN) member countries which effort focused on the human resources development through education, research and community development activities in food and nutrition area. Evidence on the effectiveness of the NGTS as the flagship program of the institution is needed to advocate the implementation of the program nationally and even regionally among the ASEAN member countries.

A cluster randomized controlled pilot trial among secondary school in Jakarta, Indonesia. The school-based nutrition intervention which consisted of multi-components could be regarded as a complex health intervention. Therefore, evaluation of its effectiveness follows the steps suggested by the UK Medical Research Council (MRC) whom devised a four-phase framework for developing and evaluating RCT's of complex interventions. This pilot trial is the 2nd phase of the framework, which will be guided by the result of the program evaluation, and aimed to assess the adherence to the whole NGTS package, determine intra-cluster correlation coefficients and effect estimates. This stage is important to inform sample size calculations for future definitive trials designed to assess the effectiveness and cost-effectiveness of a full-scale intervention as currently high-quality controlled trial on school-based health intervention in Indonesia is still lacking.

Study population is adolescents (grade 10-11; 15-17 years old) in Jakarta from ten schools (five intervention and five control);each school consisted of at least 100 students. To accommodate the Indonesian school system in urban areas, we will intentionally select schools from Jakarta Provinces, which cover 5 different municipalities, North Jakarta, East Jakarta, South Jakarta, Central Jakarta, and West Jakarta. First, recruitment will be based on the discussion with the local education office at the provincial level and ask for a list of schools considering eligibility criteria, such as having a school canteen, implementing the School Health Program (Usaha Kesehatan Sekolah/UKS), and having potential land to be utilized as a school garden. Two schools in each municipality with comparable characteristics will be selected, and then each pair will be randomized to become either the intervention or the control group. Second, selected schools will be invited to participate in the study. The intervention group will receive baseline educational intervention (Nutrition Education Capacity Building for Teachers and Management) and all components of the NGTS program. While the control group will receive only the baseline educational intervention. The baseline educational intervention will be conducted in 5 days through face-to-face delivery training mode.

The sample size for this study was determined using the formula from Hayes R and Bennett S (1999). Determination of the calculation of the main parameter assessed was based on a prior study in Ecuador of a school-based intervention to improve dietary intake outcomes, the proportion of breakfast intake. Randomization was based on the number of clusters with a total of 10 schools, considering the significant level (α) of 0.05, the coefficient of variation between groups (Intra Class Correlation/ICC) of 0.15, the power of study (β) of 80%, the ratio of cases and controls (k = 1), and the anticipated dropout of 10%. Based on the sample calculation, the number of samples per intervention group and control group was 486 people each, which was increased to 500 people. So that the total sample needed is 1,000 people, with each school consisting of 100 students.

ELIGIBILITY:
Inclusion Criteria:

* High school students in grades 10-11
* Aged 15-17 years
* Attending school in Jakarta

Exclusion Criteria:

* unwilling and/or unable to complete the questionnaire thoroughly

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge on healthy diet among children - clinical outcome | at baseline and 6 months
  Multiple choices' questionnaire
  Analyzed as Comparison of score (mean difference [MD] and 95% CI):
  * before and after the intervention
  * between the intervention and control schools
Eating attitude-clinical outcome | at baseline and 6 months
  The Eating Attitudes Test (EAT-26)
  Analyzed for a comparison of proportion eating disorder (difference and 95% CI):
  * before and after the intervention
  * between the intervention and control schools
Healthy diet behaviour-clinical outcome | at baseline and 6 months
  Fruits and vegetables, energy-dense nutrient poor food and sugary beverages consumption using semi-quantitative food frequency questionnaire (FFQ)
  Analyzed for a comparison of proportion (difference and 95% CI):
  * before and after the intervention
  * between the intervention and control schools
Physical activity-clinical outcome | at baseline and 6 months
  Rapid Assessment of Physical Activities (RAPA)
  Comparison of proportion (difference and 95% CI):
  * before and after the intervention
  * between the intervention and control schools
Nutritional status-clinical outcome | at baseline and 6 months
  Body Mass Index (BMI) for Age
mid-upper arm circumference (MUAC) | at baseline and 6 months
  Nutritional status-clinical outcome
waist circumference | at baseline and 6 months
  Nutritional status-clinical outcome

SECONDARY OUTCOMES:
School readiness on the implementation of the program - - Descriptive, Quantitative (proportion), Qualitative | Baseline
  Data source : School readiness questionnaire (Likert scale; validated)
Attendance of teachers to training sessions-proportion | at the end of the three days training
  Data source: Training attendance list
Activity report completed-proportion | during the 6-month of intervention
  Data source: NGTS monitoring dashboard
Adherence to NGTS protocol - Descriptive, Quantitative (proportion), Qualitative | during the 6-month intervention
  Data source: NGTS monitoring dashboard, interview, and observation by the field coordinator
Students' and teachers' preference and acceptance on IEC material/modules - Qualitative | during the 6-month intervention
  Data source: FGD's guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Indah S Widyahening, Professor, Principal Investigator — SEAMEO RECFON
Locations (1):
- Seameo Recfon, Jakarta, The Special Capital Region of Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Institute of Health Research and Development. Basic Health Research 2013. Jakarta: Ministry of Health of the Republic of Indonesia, National Institute of Health Research and Development; 2013.
- [Background] National Institute of Health Research and Development. Basic Health Research 2018. Jakarta: Ministry of Health of the Republic of Indonesia, National Institute of Health Research and Development; 2018.
- [Background] Glanz K, Lankenau B, Foerster S, Temple S, Mullis R, Schmid T. Environmental and policy approaches to cardiovascular disease prevention through nutrition: opportunities for state and local action. Health Educ Q. 1995 Nov;22(4):512-27. doi: 10.1177/109019819502200408. PMID 8550374
- [Background] World Health Organization. School Policy Framework: implementation of the WHO global strategy on diet, physical activity and health. Geneva: World Health Organization; 2008.
- [Background] World Health Organization. Global status report of noncommunicable diseases 2014. Geneva, Switzerland: World Health Organization; 2014.
- [Background] Parcel GS, Simons-Morton B, O'Hara NM, Baranowski T, Wilson B. School promotion of healthful diet and physical activity: impact on learning outcomes and self-reported behavior. Health Educ Q. 1989 Summer;16(2):181-99. doi: 10.1177/109019818901600204. PMID 2732062
- [Background] Silveira JA, Taddei JA, Guerra PH, Nobre MR. Effectiveness of school-based nutrition education interventions to prevent and reduce excessive weight gain in children and adolescents: a systematic review. J Pediatr (Rio J). 2011 Sep-Oct;87(5):382-92. doi: 10.2223/JPED.2123. English, Portuguese. PMID 22012577
- [Background] Verrotti A, Penta L, Zenzeri L, Agostinelli S, De Feo P. Childhood obesity: prevention and strategies of intervention. A systematic review of school-based interventions in primary schools. J Endocrinol Invest. 2014 Dec;37(12):1155-64. doi: 10.1007/s40618-014-0153-y. Epub 2014 Sep 9. PMID 25200996
- [Background] Black AP, D'Onise K, McDermott R, Vally H, O'Dea K. How effective are family-based and institutional nutrition interventions in improving children's diet and health? A systematic review. BMC Public Health. 2017 Oct 17;17(1):818. doi: 10.1186/s12889-017-4795-5. PMID 29041899
- [Background] Aloia CR, Shockey TA, Nahar VK, Knight KB. Pertinence of the recent school-based nutrition interventions targeting fruit and vegetable consumption in the United States:a systematic review. Health Promot Perspect. 2016 Mar 31;6(1):1-9. doi: 10.15171/hpp.2016.01. eCollection 2016. PMID 27123430
- [Background] Colley P, Myer B, Seabrook J, Gilliland J. The Impact of Canadian School Food Programs on Children's Nutrition and Health: A Systematic Review. Can J Diet Pract Res. 2019 Jun 1;80(2):79-86. doi: 10.3148/cjdpr-2018-037. Epub 2018 Nov 15. PMID 30430855
- [Background] Kong K, Liu J, Tao Y. Limitations of studies on school-based nutrition education interventions for obesity in China: a systematic review and meta-analysis. Asia Pac J Clin Nutr. 2016;25(3):589-601. doi: 10.6133/apjcn.092015.19. PMID 27440695
- [Background] Campbell M, Fitzpatrick R, Haines A, Kinmonth AL, Sandercock P, Spiegelhalter D, Tyrer P. Framework for design and evaluation of complex interventions to improve health. BMJ. 2000 Sep 16;321(7262):694-6. doi: 10.1136/bmj.321.7262.694. No abstract available. PMID 10987780
- [Background] Liu Z, Wu Y, Niu WY, Feng X, Lin Y, Gao A, Zhang F, Fang H, Gao P, Li HJ, Wang H; study team for the DECIDE-children study. A school-based, multi-faceted health promotion programme to prevent obesity among children: protocol of a cluster-randomised controlled trial (the DECIDE-Children study). BMJ Open. 2019 Nov 2;9(11):e027902. doi: 10.1136/bmjopen-2018-027902. PMID 31678935
- [Background] Octaria Y, Apriningsih A, Dwiriani CM, Februhartanty J. School readiness to adopt a school-based adolescent nutrition intervention in urban Indonesia. Public Health Nutr. 2021 Jun;24(S2):s72-s83. doi: 10.1017/S1368980020001299. Epub 2020 May 7. PMID 32375906
- [Background] Maehara M, Rah JH, Roshita A, Suryantan J, Rachmadewi A, Izwardy D. Patterns and risk factors of double burden of malnutrition among adolescent girls and boys in Indonesia. PLoS One. 2019 Aug 20;14(8):e0221273. doi: 10.1371/journal.pone.0221273. eCollection 2019. PMID 31430324
- [Background] Topolski TD, LoGerfo J, Patrick DL, Williams B, Walwick J, Patrick MB. The Rapid Assessment of Physical Activity (RAPA) among older adults. Prev Chronic Dis. 2006 Oct;3(4):A118. Epub 2006 Sep 15. PMID 16978493
- See also: South-east Asian Ministers of Education Organization - Regional Center for Food and Nutrition. Nutrition Goes to School Jakarta2020 — http://www.seameo-recfon.org/nutrition-goes-to-school/